CLINICAL TRIAL: NCT02578342
Title: Brain Activity and Functional Connectivity in Adults With Attention-Deficit Hyperactivity Disorder (ADHD) During Tasks of Motor Inhibition and Cognitive Switching
Brief Title: Brain Activity in Adults With ADHD During Neuropsychological Tasks
Status: Completed | Type: Observational
Sponsor: Kantonsspital Aarau (Other)
Responsible Party: Principal Investigator, Luca Remonda, Prof. Dr. med., Kantonsspital Aarau
Other Study IDs: 1410.000.055
Record Dates: First submitted 2015-08-03; First posted 2015-10-16 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Healthy volunteers: healthy volunteer between age of 20 to 55 will undergo MRI examination.
  Interventions: Device: MRI
- ADHD subjects without medication: Medication-naive subjects with ADHD (20-55 years) will undergo MRI examination.
  Interventions: Device: MRI
- ADHD subjects with medication: Subjects with ADHD (20-55 years), under medication will undergo MRI examination.
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Functional Magnetic Resonance Imaging technique measures brain activity by detecting associated changes in blood oxygenation level dependency

SUMMARY:
The aim of the study is to investigate the response on cognitive testing of healthy persons compared to adults with or without medication against ADHD.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder (ADHD) is one of the most prevalent psychiatric disorders in children and adolescents. It is characterized by inattentive, hyperactive, impulsive behaviour and neuropsychological deficits. In 40-60% of cases emerge in childhood and persists into adulthood.

The aim of the study is to investigate the response on cognitive testing of healthy persons compared to adults with or without medication against ADHD. As a secondary endpoint a more robust diagnosing method combining advanced imaging methods with neuropsychological evaluation is tested.

Neuropsychological testing, functional MRI and spectroscopy will be performed. Statistical analysis will assess differences in the functional magnetic resonance imaging, spectroscopy and neuropsychological evaluation results between three groups: 1) group of healthy volunteers, 2) participants with ADHD with medication and 3) participants with ADHD without medication.

ELIGIBILITY:
Inclusion Criteria:

* Participant is between 20-55 years old
* Participant is not pregnant

Exclusion Criteria:

* Participant is not able to consent him/herself
* Suspected or proven pregnancy
* Nursing
* Neurological diseases that could interfere with a diagnosis of ADHD
* Psychiatric comorbidity under treatment
* Previous history of psychiatric medication
* Substance abuse
* Intelligence quotient<75
* Claustrophobia
* Electrical simulator nerve or bone
* Implanted medication infusion pump
* Cerebral aneurysm clips
* Unstable medical condition

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Three groups:
  1. healthy volunteers
  2. ADHD subjects receiving medications
  3. medication-naive ADHD subjects
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-08; Primary Completion 2020-05 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Changes in blood oxygenation level dependency (BOLD) | 2 hours
  The study consist solely of one MRI examination performed within 2 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Aarau, Aarau, Canton of Aargau, Switzerland

REFERENCES:
- [Derived] Berberat J, Huggenberger R, Montali M, Gruber P, Pircher A, Lovblad KO, Killer HE, Remonda L. Brain activation patterns in medicated versus medication-naive adults with attention-deficit hyperactivity disorder during fMRI tasks of motor inhibition and cognitive switching. BMC Med Imaging. 2021 Mar 19;21(1):53. doi: 10.1186/s12880-021-00579-3. PMID 33740903